CLINICAL TRIAL: NCT04491357
Title: The Use of Prophylactic Infusion of Calcium Gluconate Compared to Placebo in Reducing the Rate of Hypocalcaemia After Total Thyroidectomy: A Double-Blinded, Randomized Controlled Trial
Brief Title: Prophylactic Infusion of Calcium Gluconate Reducing the Rate of Hypocalcaemia After Total Thyroidectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Khoo Kah Seng, Surgical Resident, Department of Surgery, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020225-8316
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Hypocalcemia
Keywords: Hypocalcaemia; Total thyroidectomy; Calcium gluconate
MeSH Terms: conditions — Hypocalcemia | interventions — Calcium Gluconate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Intervention arm will receive 1 ampoule of intravenous calcium gluconate within 4 hours of skin closure post total thyroidectomy
  Interventions: Drug: Calcium Gluconate
- Placebo arm (Placebo Comparator): Placebo arm will receive 100ml of normal saline within 4 hours of skin closure post total thyroidectomy
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Calcium Gluconate — Intravenous calcium gluconate within 4 hours of skin closure after total thyroidectomy
  Other Names: Intravenous calcium gluconate
  Arms: Intervention arm
Drug: Normal saline — Normal saline within 4 hours of skin closure after total thyroidectomy
  Arms: Placebo arm

SUMMARY:
Post-total thyroidectomy hypocalcaemia is a common complication with the rate ranging from 13-49% in a meta-analysis. However, the rate in UMMC in 2018 and 2019 were 40% and 23% respectively. It lead to prolonged hospital stay and patient dissatisfaction in the event of hypocalcaemia.

Research question: Does prophylactic intravenous calcium infusion reduces the rate of post-total thyroidectomy hypocalcaemia? This study will conduct in UMMC endocrine surgery unit with the target population who scheduled for total thyroidectomy in UMMC between 1/6/2020-1/6/2022.

After obtaining consent from participants, they will be randomised into intervention and placebo group with the ratio of 1:1. Intervention group will receive the intravenous calcium gluconate infusion and placebo group will receive saline infusion within 4 hour of skin closure. Both groups will have their serum calcium measure at 6,12,24,36,48-hour mark post surgery. Both groups will receive same oral calcium supplements.

DETAILED DESCRIPTION:
All participating patients will be randomised into intervention and placebo arm with 1:1 ratio. Intervention group will receive 1 ampoule of intravenous calcium gluconate within 4 hours of post total thyroidectomy, whereas the placebo group will received 100ml of normal saline only. Both groups will receive same oral calcium supplements post surgery. Both groups will have their serum calcium measure at 6,12,24,36,48-hour mark post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years old
* Scheduled for total thyroidectomy in UMMC

Exclusion Criteria:

* Their age outside the range of 18-80
* Have parathyroid disorders or end stage renal failure
* On calcium or vitamin D supplements prior to surgery
* Have deranged calcium homeostasis (outside the normal range of 2.2-2.6 mmol/L)
* Scheduled for total thyroidectomy plus lymph node dissection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of hypocalcaemia after total thyroidectomy | first 48 hours after total thyroidectomy
  To determine whether prophylactic infusion of calcium gluconate reduces the rate of hypocalcaemia after total thyroidectomy compared to placebo treatment

SECONDARY OUTCOMES:
Length of hospital stay | first 48 hours after total thyroidectomy
  To determine whether prophylactic infusion of calcium gluconate reduces the length of hospital stay compared to placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Kah Seng Khoo, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Not to share IPD to other researchers

REFERENCES:
- [Derived] Khoo KS, Yeo A, Mirzan Asfian MRB, Ng KL. The use of prophylactic infusion of calcium gluconate compared to placebo in reducing the rate of early hypocalcaemia after total thyroidectomy: a double-blinded, randomized controlled trial. Gland Surg. 2024 Aug 31;13(8):1378-1386. doi: 10.21037/gs-24-190. Epub 2024 Aug 28. PMID 39282041